CLINICAL TRIAL: NCT00691262
Title: A Long Term, Non-comparative, Multi-centre Study to Further Evaluate the Response to Treatment and Safety of 0.03% Tacrolimus Ointment Administered in Pediatric Patients With Moderate to Severe Atopic Dermatitis.
Brief Title: Study to Evaluate the Response to Treatment and Safety of 0.03% Tacrolimus (FK506) Ointment Administered in Pediatric Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-06-IT-02
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatitis; Prograf; Tacrolimus; FK506; Tacrolimus ointment
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment

INTERVENTIONS:
Drug: tacrolimus ointment — transdermal
  Other Names: FK506

SUMMARY:
Objective of this study is to further assess the response to treatment and safety of 0.03% tacrolimus (FK506) ointment when used for 6 months in pediatric patients with moderate to severe atopic dermatitis, known to be responsive to topical steroids.

DETAILED DESCRIPTION:
The main phase is 6 month duration, but the follow-up phase up to 12 months will allow the collection of RTT and safety data in a period which will include all seasons in each patient, to account for seasonal variability which strongly affect AD course.

ELIGIBILITY:
Inclusion Criteria:

* Patient may be male or female of any ethnic group
* Patient is aged 2 years to 15 years (not having completed his/her 16th birthday) and suffers from moderate to severe atopic dermatitis (Rajka/Langeland score of at least 4.5).
* Patient known to be responsive to topical steroids
* Patient's legal representative has given written informed consent. If the patient is capable of understanding the purposes and risks of the trial written informed consent has been obtained from the patient as well. Female patients of childbearing potential must agree to maintain adequate birth control practice during the trial period and during the first four weeks after the end of the study
* Patient meets the following wash-out criteria:

  * Topical corticosteroids
  * Systemic corticosteroids (for the treatment of AD only)
  * Systemic non-steroidal immunosuppressants (e.g. cyclosporine, methotrexate)
  * Other investigational drugs
  * Light Treatments (UVA, UVB)
* Patient has not taken/patient and legal representative agree that the patient does not take for the complete study period any medication or therapy prohibited by the protocol

Exclusion Criteria:

* Patient has a genetic epidermal barrier defect such as Netherton's syndrome or generalised erythroderma
* Patient is pregnant or breast-feeding
* Patient has a skin infection on the affected (and to be treated) area
* Patient has a known hypersensitivity to macrolides in general, to Tacrolimus or any excipient of the ointment
* Patient is simultaneously participating in any other drug trial or less than 28 days have passed between the end of the previous trial and this one
* Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder or condition which, in the opinion of the investigator, may invalidate the communication with the investigator
* Patient is known to be HIV positive

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The rate of patients with at least 50% (i.e. at least moderate) improvement according to the physician's global evaluation of clinical response at month 6/end of study (if before month 6) visit | 1 year

SECONDARY OUTCOMES:
The rate of patients with at least 50% (i.e. at least moderate) improvement according to the physician's global evaluation of clinical response at month 12/end of study (if before month 6) visit | 1 year
The rate of patients with at least 60% improvement in the Score in Atopic Dermatitis (SCORAD) at month 6/end of study (if before month 6) visit and at month 12/end of study (if after month 6) visit, each compared to baseline (day 1) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (7):
- Italy (7):
  - Bologna
  - Catania
  - Genova
  - Lecco
  - Napoli
  - Padua
  - Roma